CLINICAL TRIAL: NCT01015443
Title: A Multi-national, Double-blind, Placebo-controlled, Randomized, Phase III Clinical Trial of the Cancer Vaccine Stimuvax® (L-BLP25 or BLP25 Liposome Vaccine) in Asian Subjects With Stage III, Unresectable, Non-small Cell Lung Cancer (NSCLC) Who Have Demonstrated Either Stable Disease or Objective Response Following Primary Chemo-radiotherapy
Brief Title: Cancer Vaccine Study for Stage III, Unresectable, Non-small Cell Lung Cancer (NSCLC) in the Asian Population
Acronym: INSPIRE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study is terminated prematurely as the sponsor decided to discontinue program with Tecemotide in NSCLC.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMR63325-012
Record Dates: First submitted 2009-10-01; First posted 2009-11-18 (Estimated); Results first posted 2016-08-02 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Carcinoma; Tecemotide; L-BLP25; Cyclophosphamide; placebo controlled; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — L-BLP25; Single Person; Cyclophosphamide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Investigational Arm (Experimental): Tecemotide (L-BLP25) + Single low dose cyclophosphamide + Best supportive care (BSC)
  Interventions: Biological: Tecemotide; Drug: Single low dose cyclophosphamide; Other: Best Supportive Care (BSC)
- Control Arm (Placebo Comparator): Saline + Placebo + Best supportive care (BSC)
  Interventions: Drug: Placebo; Other: Saline; Other: Best Supportive Care (BSC)

INTERVENTIONS:
Biological: Tecemotide — Subjects will receive 8 consecutive weekly subcutaneous vaccinations with 918 microgram (mcg) of tecemotide (L-BLP25) at Week 1, 2, 3, 4, 5, 6, 7, and 8 (primary treatment phase) and then at 6-Week intervals, beginning at Week 14 (maintenance phase) until disease progression (PD) is documented or the subject discontinues for any other reason.
  Other Names: L-BLP25; Stimuvax
  Arms: Investigational Arm
Drug: Single low dose cyclophosphamide — A single intravenous (IV) infusion of 300 milligram per square meter (mg/m^2) (to a maximum 600 mg) of cyclophosphamide will be given 3 days before the first administration of tecemotide.
  Arms: Investigational Arm
Drug: Placebo — Subjects will receive 8 consecutive weekly subcutaneous vaccinations of tecemotide (L-BLP25) matching placebo at Week 1, 2, 3, 4, 5, 6, 7 and 8 followed by maintenance treatment at 6-Week intervals, beginning at Week 14, until PD is documented or the subject discontinues for any other reason.
  Arms: Control Arm
Other: Saline — A single IV infusion of 0.9 percent (%) sodium chloride (saline) will be given 3 days before first placebo vaccination.
  Arms: Control Arm
Other: Best Supportive Care (BSC) — The BSC will be provided as per the investigator's discretion, and is not limited to palliative radiation, psychosocial support, analgesics and nutritional support.

SUMMARY:
The purpose of this study is to determine whether the cancer vaccine tecemotide (L-BLP25) in addition to best supportive care is effective in prolonging the lives of Asian subjects with unresectable stage III non-small cell lung cancer in comparison to a placebo plus best supportive care (a so-called placebo controlled study).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented unresectable stage III non-small cell lung cancer (NSCLC)
* Documented stable disease or objective response, according to Response Evaluation Criteria In Solid Tumors Version 1.0 (RECIST v1.0) after primary concomitant chemo-radiotherapy for unresectable stage III disease, within four weeks (28 days) prior to randomization
* Receipt of concomitant chemo-radiotherapy. The chemotherapy-part must have been platinum-based, must have been administered with a minimum of two cycles overlap with radiotherapy (one cycle lasts either 3 or 4 weeks depending on the chemotherapy regimen), and a minimum of two platinum-based chemotherapy administrations must have been given during radiotherapy. Purely radio sensitizing doses of chemotherapy are not acceptable. Radiotherapy must have delivered a radiation dose of >= (greater than or equal to) 50 Gray (Gy). Induction or consolidation chemotherapy is allowed and if given, should be accounted as part of primary thoracic chemoradiotherapy. Subjects must have completed the primary thoracic chemo-radiotherapy at least four weeks (28 days) and no later than 12 weeks (84 days) prior to randomization. Subjects who received prophylactic brain irradiation as part of primary chemo-radiotherapy are eligible
* Geographically accessible for ongoing follow-up, and committed to comply with the designated visits
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* A platelet count >= the lower limit of normal for the site or >= 100 x 10^9 per liter (/Liter) (whichever is greater); white blood cell (WBC) >= 2.5 x 10^9/Liter and haemoglobin >= 90 gram per liter (g/L)
* >=18 years of age (or minimum age of legal consent consistent with local regulations, if minimum is greater than [>] 18 years of age)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

Pre-Therapies*:

* Prior sequential chemo-radiotherapy
* Lung-cancer-specific therapy (including surgery) other than primary chemoradiotherapy
* Immunotherapy (e.g., interferons, tumor necrosis factor [TNF], interleukins, or biological response modifiers [granulocyte macrophage colony stimulating factor {GMCSF}, granulocyte colony stimulating factor {G-CSF}, macrophage-colony stimulating factor {M-CSF}], monoclonal antibodies) within four weeks (28 days) prior to randomization
* Investigational systemic drugs (including off-label use of approved products) within four weeks (28 days) prior to randomization

Disease Status:

* Metastatic disease
* Malignant pleural effusion at initial diagnosis and/or at trial entry
* Past or current history of neoplasm other than lung carcinoma, except for curatively treated non-melanoma skin cancer, in situ carcinoma of the cervix, or other cancer curatively treated and with no evidence of disease for at least 5 years
* Autoimmune disease
* A recognized immunodeficiency disease including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia; subjects who have hereditary or congenital immunodeficiencies
* Any preexisting medical condition requiring chronic steroid or immunosuppressive therapy (steroids for the treatment of radiation pneumonitis are allowed)
* Known active Hepatitis B infection and/or Hepatitis C infection
* Signs and symptoms suggestive of transmissible spongiform encephalopathy, or of family members who suffer(ed) from such

Physiological Functions:

* Clinically significant hepatic dysfunction
* Clinically significant renal dysfunction
* Clinically significant cardiac disease
* Splenectomy
* Infectious process that in the opinion of the investigator could compromise the subject's ability to mount an immune response

Standard Safety:

* Pregnant or breastfeeding women, women of childbearing potential, unless using effective contraception as determined by the investigator
* Known drug abuse or alcohol abuse
* Participation in another clinical trial (excluding purely observational studies) within the past 28 days
* Requires concurrent treatment with a non-permitted drug
* Known hypersensitivity to any of the trial treatment ingredients
* Legal incapacity or limited legal capacity
* Any other reason that, in the opinion of the investigator precludes the subject from participating in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2009-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical responsible, Study Director — Merck Serono (Beijing), Pharmaceutical R&D Co., Ltd., an Affiliate of Merck KGaA Darmstadt, Germany
Locations (47):
- China (29):
  - 307 Hospital of Chinese PLA, Beijing
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital, Beijing
  - Cancer Institue & Hospital, Chinese Academy of Medical Sciences, Beijing
  - The First Hospital of Jilin University, Changchun
  - Jillin Provincial Cancer Hospital, Changchun
  - West China Hospital of Sichuan University, Chengdu, Sichuan Province
  - Southwest Hospital of the Third Military Medical University, Chongqing
  - The Second Affiliate Hospital of the Third Military Medical University, Chongqing
  - Fujian Province Tumor Hospital, Fuzhou
  - Guangdong General Hospital, Guangzhou
  - The First Affilated Hospital of Guangzhou Medical College, Guangzhou
  - Heilongjiang Cancer Hospital, Haerbin
  - China PLA General Hospital, Haidian Districk, Beijing
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Yunan Tumor Hospital, Kunming
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - PLA 81 Hospital, Nanjing
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Fundan University Cancer Hospital, Shanghai
  - Shangahi Pulmonary Hosptial, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Shanghai Chest Hosptial, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - Tongji Hospital of Tongji Medical Colleague of Huazhong University of Science and Technology, Wuhan
  - Peking Union Medical College Hospital, XiCheng District, Beijing
  - Subei People's Hospital, Yangzhou
- Hong Kong (4):
  - Queen Elizabeth Hospital, Kowloon
  - Tuen Mun Hospital, New Territories
  - Queen Mary Hospital, Pok Fu Lam
  - Prince of Wales Hospital, Shatin, N.T.
- National University Hospital, Singapore, Singapore
- South Korea (4):
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsi University College of Medicine, Seoul
  - St. Mary's Hospital, The Catholic University of Korea, Seoul
- Taiwan (9):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation, Kaohsiung, Kaohsiung County
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital, Liouying, Tainan County
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Dept of Chest, Taipei
  - Chang Gung medical Foundation, Linkou Branch, Taoyuan District

REFERENCES:
- [Derived] Zhu J, Yuan Y, Wan X, Yin D, Li R, Chen W, Suo C, Song H. Immunotherapy (excluding checkpoint inhibitors) for stage I to III non-small cell lung cancer treated with surgery or radiotherapy with curative intent. Cochrane Database Syst Rev. 2021 Dec 6;12(12):CD011300. doi: 10.1002/14651858.CD011300.pub3. PMID 34870327
- [Derived] Wu YL, Park K, Soo RA, Sun Y, Tyroller K, Wages D, Ely G, Yang JC, Mok T. INSPIRE: A phase III study of the BLP25 liposome vaccine (L-BLP25) in Asian patients with unresectable stage III non-small cell lung cancer. BMC Cancer. 2011 Oct 7;11:430. doi: 10.1186/1471-2407-11-430. PMID 21982342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject (informed consent): 03 Dec 2009/10-Sep-2014. Data cut-off date: June 2015; Subjects were randomized at 45 centers in 5 countries worldwide.
Pre-assignment Details: A total of 350 subjects were screened for eligibility and 285 subjects were enrolled and randomized.
Groups:
- Tecemotide (L-BLP25)+Cyclophosphamide+Best Supportive Care: A single intravenous (IV) infusion of 300 milligram per square meter (mg/m^2) (to a maximum 600 mg) of low dose cyclophosphamide was given 3 days prior to first tecemotide (L-BLP25) vaccination. After receiving single low dose cyclophosphamide, subjects received 8 consecutive weekly (Week 1, 2, 3, 4, 5, 6, 7, and 8 primary treatment phase) subcutaneous tecemotide (L-BLP25) vaccinations at a dose of 918 microgram (mcg) and then at 6-Week interval, beginning at Week 14 (maintenance phase) until disease progression (PD) is documented or the subject discontinued for any other reason. The best supportive care (BSC) was provided as per the investigator's discretion and was not limited to palliative radiation, psychosocial support, analgesics and nutritional support.
- Saline + Placebo + BSC: A single IV infusion of 0.9 percent (%) sodium chloride (saline) was administered 3 days prior to first placebo vaccination. After receiving saline solution, subjects received 8 consecutive weekly subcutaneous vaccinations with placebo at Week 1, 2, 3, 4, 5, 6, 7 and 8 followed by maintenance treatment at 6-Week intervals, beginning at Week 14, until PD is documented or the subject discontinued for any other reason. The BSC was provided as per the investigator's discretion and was not limited to palliative radiation, psychosocial support, analgesics and nutritional support.
Period: Overall Study
Arm/Group | Tecemotide (L-BLP25)+Cyclophosphamide+Best Supportive Care | Saline + Placebo + BSC
Started | 191 | 94
Treated | 191 | 93
Completed | 191 | 94
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention to treat (ITT) subjects included all the subjects randomized into the study.
Groups:
- Tecemotide (L-BLP25)+Cyclophosphamide+BSC: A single IV infusion of 300 mg/m^2 (to a maximum 600 mg) of low dose cyclophosphamide was given 3 days prior to first tecemotide (L-BLP25) vaccination. After receiving single low dose cyclophosphamide, subjects received 8 consecutive weekly (Week 1, 2, 3, 4, 5, 6, 7, and 8 primary treatment phase) subcutaneous tecemotide (L-BLP25) vaccinations at a dose of 918 mcg and then at 6-Week interval, beginning at Week 14 (maintenance phase) until PD is documented or the subject discontinued for any other reason. The BSC was provided as per the investigator's discretion and was not limited to palliative radiation, psychosocial support, analgesics and nutritional support.
- Saline + Placebo + BSC: A single IV infusion of 0.9% sodium chloride (saline) was administered 3 days prior to first placebo vaccination. After receiving saline solution, subjects received 8 consecutive weekly subcutaneous vaccinations with placebo at Week 1, 2, 3, 4, 5, 6, 7 and 8 followed by maintenance treatment at 6-Week intervals, beginning at Week 14, until PD is documented or the subject discontinued for any other reason. The BSC was provided as per the investigator's discretion and was not limited to palliative radiation, psychosocial support, analgesics and nutritional support.
- Total: Total of all reporting groups
Arm/Group | Tecemotide (L-BLP25)+Cyclophosphamide+BSC | Saline + Placebo + BSC | Total
Number analyzed (Participants) | 191 | 94 | 285
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (8.93) | 59.3 (9.08) | 57.4 (9.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 18 | 49
  Male | 160 | 76 | 236

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Time
Description: OS time was measured as the time (in months) between the date of randomization and the date of death. For subjects alive or lost to follow-up at time of analysis, the time between the date of randomization and the date on which the subject was last known alive was calculated and used as a censored observation in the analysis.
Time Frame: From the date of randomization until death, assessed up to 5.6 years
Population: The modified intent-to-treat (mITT) analysis set was based on the intention-to-treat (ITT) analysis set (ITT analysis set included all the subjects randomized into the study), but included only subjects with concurrent primary chemo-radiotherapy and prospectively excluded the 5 subjects who were randomized prior to the clinical hold.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tecemotide (L-BLP25)+Cyclophosphamide+BSC | Saline + Placebo + BSC
Number analyzed (Participants) | 135 | 68
Months | NA [28.7 to NA] — Fewer subjects were randomized than planned and analysis was performed earlier than planned due to termination of the tecemotide (L-BLP25) program which resulted in few events. Hence, median and upper limit of confidence interval were not estimable. | NA [23.7 to NA] — Fewer subjects were randomized than planned and analysis was performed earlier than planned due to termination of the tecemotide (L-BLP25) program which resulted in few events. Hence, median and upper limit of confidence interval were not estimable.
Statistical Analysis 1: Comparison: Tecemotide (L-BLP25)+Cyclophosphamide+BSC vs Saline + Placebo + BSC; Test type: Superiority or Other; p = 0.921, Adjusted log rank; Hazard Ratio (HR) = 1.032, 95% CI 2-sided [0.552 to 1.931]

2. Secondary Outcome: Time to Symptom Progression (TTSP)
Description: TTSP was measured from randomization to symptomatic progression by lung cancer symptom scale (LCSS) used to measure symptom changes relevant to quality of life (QoL).It consisted of 9 items focused on cancer symptoms (loss of appetite, fatigue, cough, shortness of breath, blood in sputum, pain, symptoms of cancer, illness affecting normal activity, QoL).For each symptom score distance from left boundary to point where subject has marked line was measured in millimeters (mm).Total scale length was 100 mm. Symptomatic progression was defined as increase/worsening of average symptomatic burden index (ASBI) (mean of 6 major lung cancer specific symptom scores);Worsening defined as 10% increase of scale breadth from baseline. Score 0 indicate no/minimum symptoms;100 indicates maximum level of symptoms. Subjects without symptomatic progression/lost to follow-up at time of analysis: time from date of randomization to date of last LCSS assessment was calculated & used as censored observation.
Time Frame: From the date of randomization to the date of symptomatic progression, assessed up to 5.6 years
Population: The mITT analysis set was based on the ITT analysis set (ITT analysis set included all the subjects randomized into the study), but included only subjects with concurrent primary chemo-radiotherapy and prospectively excluded the 5 subjects who were randomized prior to the clinical hold.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tecemotide (L-BLP25)+Cyclophosphamide+BSC | Saline + Placebo + BSC
Number analyzed (Participants) | 135 | 68
Months | 19.3 [16.7 to NA] — Fewer subjects were randomized than planned and analysis was performed earlier than planned due to termination of the tecemotide (L-BLP25) program which resulted in few events. Hence, upper limit of confidence interval was not estimable. | 24.2 [10.8 to NA] — Fewer subjects were randomized than planned and analysis was performed earlier than planned due to termination of the tecemotide (L-BLP25) program which resulted in few events. Hence, upper limit of confidence interval was not estimable.

3. Secondary Outcome: Time to Progression (TTP)
Description: Time from randomization to radiological confirmation of disease progression (PD) as determined by the investigator. PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions from nadir, or the appearance of one or more new lesions as per RECIST version 1.0. For subjects without radiological confirmed PD who discontinued or died due to PD, the date of trial treatment discontinuation was used as event date. Subjects who missed 2 consecutive scheduled doses without evaluable assessment for the related visits and who were lost to follow-up thereafter were considered as having PD, TTP was calculated from the date of randomization to the date of their first missed treatment. Subjects without PD at time of analysis are censored at either date of last vaccination or death or discontinuation of treatment or lost to follow-up.
Time Frame: From the date of randomization to the date of radiological confirmation of PD, assessed up to 5.6 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tecemotide (L-BLP25)+Cyclophosphamide+BSC | Saline + Placebo + BSC
Number analyzed (Participants) | 135 | 68
Months | 6.4 [5.5 to 8.6] | 7.5 [5.9 to 15.2]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Time from randomization to objective disease progression (PD) as determined by the investigator or death. PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions from nadir, or the appearance of one or more new lesions as per RECIST version 1.0. Subjects who missed 2 consecutive scheduled doses without evaluable assessment for the related visits and who were lost to follow-up thereafter were considered as having PD, and the PFS was calculated from the date of randomization to the date of their first missed treatment. PFS time for subjects without an event was censored as of the date of last performed imaging.
Time Frame: From the date of randomization to PD, assessed up to 5.6 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tecemotide (L-BLP25)+Cyclophosphamide+BSC | Saline + Placebo + BSC
Number analyzed (Participants) | 135 | 68
Months | 7.0 [5.5 to 8.7] | 8.7 [5.9 to 15.2]

5. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF was time from randomization to discontinuation of trial treatment for any reason as reported by the investigator. For subjects still receiving treatment at the time of analysis, the time between the date of randomization and the last date of treatment will be used as a censored observation in the analysis. Subjects who missed 2 consecutive scheduled doses without evaluable assessment for the related visits and who were lost to follow-up thereafter were considered treatment failure and the TTF was calculated from the date of randomization to the date of their first missed treatment.
Time Frame: From the date of randomization to the date of first missed treatment, assessed up to 5.6 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tecemotide (L-BLP25)+Cyclophosphamide+BSC | Saline + Placebo + BSC
Number analyzed (Participants) | 135 | 68
Months | 4.6 [4.5 to 6.0] | 4.6 [3.3 to 5.9]

6. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Discontinuation and TEAEs Leading to Death
Description: An Adverse Event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A Serious Adverse Event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs were defined as the AEs that occur between first dose of study drug administration and 42 days after the last dose of study drug administration that were absent before treatment or that worsened relative to pretreatment state. Number of subjects with TEAE leading to death and permanent discontinuation of any trial treatment were presented.
Time Frame: From the first dose of study drug administration until 42 days after the last dose of study drug administration, assessed up to 5.6 years
Population: Safety analysis set included all subjects who received at least one dose of trial treatment.
Measure: Number; unit: Subjects
Arm/Group | Tecemotide (L-BLP25)+Cyclophosphamide+BSC | Saline + Placebo + BSC
Number analyzed (Participants) | 191 | 93
Subjects
  TEAEs | 156 | 73
  Serious TEAE | 34 | 21
  TEAEs leading to discontinuation | 22 | 11
  TEAEs leading to death | 4 | 2

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration until 42 days after the last dose of study drug administration, assessed up to 5.6 years
Description: Safety analysis set included all subjects who received at least one dose of trial treatment.
Arm/Group | Tecemotide (L-BLP25)+Cyclophosphamide+BSC | Saline + Placebo + BSC
Serious Adverse Events (participants affected / at risk) | 34/191 | 21/93
Other Adverse Events (participants affected / at risk) | 151/191 | 70/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tecemotide (L-BLP25)+Cyclophosphamide+BSC (N=191) | Saline + Placebo + BSC (N=93)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 2 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Disease progression (General disorders) | 8 | 3
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Empyema (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Necrotising fasciitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 3
Sepsis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary radiation injury (Injury, poisoning and procedural complications) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 3 | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tecemotide (L-BLP25)+Cyclophosphamide+BSC (N=191) | Saline + Placebo + BSC (N=93)
Abdominal pain upper (Gastrointestinal disorders) | 6 | 5
Constipation (Gastrointestinal disorders) | 5 | 8
Diarrhoea (Gastrointestinal disorders) | 7 | 5
Chest discomfort (General disorders) | 5 | 6
Disease progression (General disorders) | 11 | 3
Fatigue (General disorders) | 24 | 13
Non-cardiac chest pain (General disorders) | 15 | 11
Oedema peripheral (General disorders) | 5 | 5
Pyrexia (General disorders) | 11 | 11
Upper respiratory tract infection (Infections and infestations) | 15 | 7
Radiation pneumonitis (Injury, poisoning and procedural complications) | 8 | 6
Decreased appetite (Metabolism and nutrition disorders) | 20 | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 5
Dizziness (Nervous system disorders) | 16 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 47 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 15
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Rash (Skin and subcutaneous tissue disorders) | 13 | 2

LIMITATIONS AND CAVEATS:
The study is terminated prematurely as the sponsor decided to discontinue program with Tecemotide in NSCLC.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other